CLINICAL TRIAL: NCT06912555
Title: A Randomized Study to Investigate the Effect of Low-calorie Diets With Different Macronutrient Composition and Macronutrient Distribution in Shift Workers With Prediabetes or Type 2 Diabetes and Overweight or Obesity.
Brief Title: Effect of Low-calorie Diets With Different Macronutrient Composition and Macronutrient Distribution in Shift Workers With Prediabetes or Type 2 Diabetes and Overweight or Obesity.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Principal Investigator, Rocio Mateo-Gallego, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PI23/558
Record Dates: First submitted 2025-03-24; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Overweight or Obesity; PreDiabetes
Keywords: shift work; hight protein diet
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Prediabetic State | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A. Low-calorie and high-protein diet with high-protein dinner (60% of total daily protein) (Experimental): The macronutrient distribution will be initially based on a protein intake of 1.3-1.5 g/kg of body weight. From this protein intake, the total calorie intake will be calculated, and 30% of these calories will be allocated to fat consumption. The remaining calories will be allocated to carbohydrate consumption, depending on the amount of protein consumed.
  The protein will be distributed as follows: breakfast and lunch (~40%), and dinner (~60%).
  The caloric restriction will be moderate, involving a reduction of 30% of the total energy expenditure, specifically calculated for each individual. This reduction will result in approximately 400-600 kcal decrease per day compared to the participant's usual energy needs. It is important to note that the caloric content of the diet will never be less than 1200 kcal per day, as such a diet may not meet the participant's nutritional requirements.
  Interventions: Other: Diet
- B. Low-calorie and high-protein diet with low-protein dinner (15% of total daily protein) (Experimental): The macronutrient distribution will be initially based on a protein intake of 1.3-1.5 g/kg of body weight. From this protein intake, the total calorie intake will be calculated, and 30% of these calories will be allocated to fat consumption. The remaining calories will be allocated to carbohydrate consumption, depending on the amount of protein consumed.The protein will be distributed as follows: breakfast and lunch (~85%), and dinner (~15%).
  The caloric restriction will be moderate, involving a reduction of 30% of the total energy expenditure, specifically calculated for each individual. This reduction will result in approximately 400-600 kcal decrease per day compared to the participant's usual energy needs. It is important to note that the caloric content of the diet will never be less than 1200 kcal per day, as such a diet may not meet the participant's nutritional requirements.
  Interventions: Other: Diet
- C. Low-calorie and regular-protein diet (Experimental): The macronutrient distribution will be initially based on a protein intake of 0.8 g/kg of body weight. From this protein intake, the total calorie intake will be calculated, and 30% of these calories will be allocated to fat consumption. The remaining calories will be allocated to carbohydrate consumption, depending on the amount of protein consumed.
  The caloric restriction will be moderate, involving a reduction of 30% of the total energy expenditure, specifically calculated for each individual. This reduction will result in approximately 400-600 kcal decrease per day compared to the participant's usual energy needs. It is important to note that the caloric content of the diet will never be less than 1200 kcal per day, as such a diet may not meet the participant's nutritional requirements.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — The nutritional plan will be initially based on a protein intake of 1.3 to 1.5 g per kilogram of body weight. From this, the total daily calorie intake is calculated, with 30% of the calories allocated to fats. The remaining calories will be assigned to carbohydrates, depending on the protein intake. Protein distribution will be approximately 40% at breakfast and lunch, and 60% at dinner. Caloric restriction will be moderate, reducing the total energy expenditure by 30%-calculated individually-which translates to an approximate decrease of 400 to 600 kcal per day compared to the participant's usual energy needs. It is important to note that the diet will never provide less than 1200 kcal per day to ensure that the minimum nutritional requirements are met.
  Arms: A. Low-calorie and high-protein diet with high-protein dinner (60% of total daily protein)
Other: Diet — The macronutrient plan will include a protein intake of 1.3 to 1.5 g per kilogram of body weight. Based on this protein amount, the total daily caloric intake will be determined, allocating 30% of the calories to fat consumption. The remaining calories will be assigned to carbohydrates, proportional to the protein intake. Protein distribution will be approximately 85% during breakfast and lunch and 15% at dinner. The caloric restriction will be moderate, with a 30% reduction in total energy expenditure calculated individually, resulting in an approximate decrease of 400 to 600 kcal per day compared to the participant's usual energy needs. It is important to note that the diet will never contain fewer than 1200 kcal per day, ensuring that the participant's nutritional requirements are met.
  Arms: B. Low-calorie and high-protein diet with low-protein dinner (15% of total daily protein)
Other: Diet — The macronutrient plan will include a protein intake of 0.8 g per kilogram of body weight. From this protein amount, the total daily calorie intake will be calculated, with 30% of the calories allocated to fats. The remaining calories will be assigned to carbohydrates, depending on the protein intake. Caloric restriction will be moderate, reducing the total energy expenditure by 30%-calculated individually-which translates to an approximate decrease of 400 to 600 kcal per day compared to the participant's usual energy needs. It is important to note that the diet will never contain fewer than 1200 kcal per day, ensuring that the participant's nutritional requirements are met.
  Arms: C. Low-calorie and regular-protein diet

SUMMARY:
Background and Aims: Shift work, particularly involving night shifts, is associated with increased risk of metabolic disturbances such as type 2 diabetes mellitus (T2DM). Thus, it is important to explore mechanisms underlying this deleteroius effect and strategies that could prevent or mitigate it. The aim of the study is to investigate the effect of three low-calorie diets with different macronutrients composition and distribution along day on glucose metabolism and other health outcomes in overweight or obese shift workers with prediabetes or T2DM.

Methods: In this randomized controlled trial, 120 shift workers with a BMI > 27.5 kg/m2 and diagnosed with prediabetes or T2DM will be recruited. The trial assesses three low-calorie diets effects on glucose metabolism, body composition, and health outcomes over 12 weeks. These diets include: A) high-protein dinner (60% of total daily protein), B) low-protein dinner (15% of total daily protein), and C) normoproteic diet.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ranging between 27.5 and 40 kg/m2.
* Presence of prediabetes (fasting glucose between 100-125 mg/dL and/or glycated hemoglobin between 5.7 and 6.4%) or type 2 diabetes mellitus (fasting glucose ≥ 126 mg/dL and/or glycated hemoglobin ≥ 6.5% and/or currently taking metformin), based on the criteria of the American Diabetes Association.
* Engaged in shift work, including night shifts, for at least 1 year and intending to maintain this schedule in the upcoming months.
* Provide written informed consent for voluntary participation in the study after reviewing the participant information sheet and addressing any resulting queries.

Exclusion Criteria:

* Treatment with antidiabetic medications (oral or subcutaneous) or insulin in the last 2 months, except for stable use of metformin or Dipeptidyl peptidase 4 (DPP-4) inhibitors for a minimum of 6 months.
* Treatment with lipid-lowering agents in an unstable manner for at least 6 months prior to study entry.
* Regular consumption of functional foods such as phytosterols or red yeast rice, which have a significant effect on lipid or glucose metabolism, in an unstable manner for at least 6 months prior to study entry.
* Presence of other chronic conditions that are not well-controlled and could interfere with study outcomes, such as cardiovascular disease, renal disease, or liver disease.
* Presence of uncontrolled endocrine disorders, including hypothyroidism.
* Use of medications that could interfere with lipid and/or glucose metabolism, unless taken stably throughout the study.
* Consumption of sleep supplements, except for stable use for 6 months with the intention to continue stable use throughout the study.
* Presence of any laboratory abnormalities that could affect study results.
* Weight gain or loss of ≥ 5% in the last 3 months.
* Use of vitamin supplements in an unstable manner for at least 6 months prior to study entry.
* High intake of alcohol (> 30 g of ethanol) on a regular basis.
* Pregnancy or intention to become pregnant during the study.
* Severe illness of any kind with a life expectancy of less than 1 year or that, in the investigators' judgment, limits uniform dietary intake throughout the study.
* Any other circumstance that, in the investigators' judgment, would impede adequate adherence to the proposed nutritional intervention (e.g., frequent travel during the study, inability to attend visits due to personal or work-related circumstances, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucose change. | After 3 months of intervention.
  Glucose change assessed by difference in fasting glucose concentration (mg/dL and %) comparing 3 months visit with respect to baseline.
Glycated hemoglobin change. | After 3 months of intervention.
  Glycated change assessed by difference in glycated hemoglobin concentration (%) comparing 3 months visit with respect to baseline.
Insulin change. | After 3 months of intervention.
  Insulin change assessed by difference in fasting insulin concentration (UI/mL and %) comparing 3 months visit with respect to baseline.
HOMA-IR change. | After 3 months of intervention.
  HOMA-IR change assessed by difference in HOMA-IR concentration (absolute units and %) comparing 3 months visit with respect to baseline.
Body fat mass change. | After 3 months of intervention.
  Body fat mass change assessed by difference in fat mass (%) comparing 3 months visit with respect to baseline.
Fat-free mass change. | After 3 months of intervention.
  Fat-free mass change assessed by difference in fat free-mass (%) comparing 3 months visit with respect to baseline.
Visceral fat mass change. | After 3 months of intervention.
  Visceral fat mass change assessed by difference in visceral fat mass (kg and %) comparing 3 months visit with respect to baseline.

SECONDARY OUTCOMES:
Total cholesterol change. | After 3 months of intervention.
  Total cholesterol change assessed by difference in fasting total cholesterol concentration (mg/dL and %) comparing 3 months visit with respect to baseline.
LDL cholesterol change. | After 3 months of intervention.
  LDL cholesterol change assessed by difference in fasting LDL cholesterol concentration (mg/dL and %) comparing 3 months visit with respect to baseline.
HDL cholesterol change. | After 3 months of intervention.
  HDL cholesterol change assessed by difference in fasting HDL cholesterol concentration (mg/dL and %) comparing 3 months visit with respect to baseline.
Triglycerides change. | After 3 months of intervention.
  Triglycerides change assessed by difference in fasting Triglycerides concentration (mg/dL and %) comparing 3 months visit with respect to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Investigación Sanitaria Aragón, Hospital Universitario Miguel Servet, Universidad de Zaragoza, Zaragoza, Spain, Spain

IPD SHARING:
Plan to Share IPD: No